CLINICAL TRIAL: NCT07247760
Title: PATIENT SATISFACTION AND MASKING OF WHITE SPOT LESIONS AFTER HOME WHITENING WITH 10% CARBAMIDE PEROXIDE: CLINICAL TRIAL
Brief Title: PATIENT SATISFACTION AND MASKING OF WHITE SPOT LESIONS AFTER HOME WHITENING WITH 10% CARBAMIDE PEROXIDE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Isabel Giráldez de Luis, PhD DDS, Universidad Rey Juan Carlos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URJC_IDIBO_5
Record Dates: First submitted 2025-11-16; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: White Spot Lesions
Keywords: white spot; bleaching; satisfaction; gingival irritation; sensitivity
MeSH Terms: conditions — Personal Satisfaction; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whitening treatment for teeth with white spot lesions (Experimental): Whitening treatment with 10% carbamide peroxide on teeth with white spot lesions. Assess patient satisfaction with the masking of white spot lesions and the occurrence of tooth sensitivity and gingival irritation.
  Interventions: Other: Whitening treatment with 10% carbamide peroxide on teeth with white spot lesions

INTERVENTIONS:
Other: Whitening treatment with 10% carbamide peroxide on teeth with white spot lesions — Whitening treatment with 10% carbamide peroxide on teeth with white spot lesions. Assess patient satisfaction with the masking of white spot lesions and the occurrence of tooth sensitivity and gingival irritation.

SUMMARY:
The clinical trial aims to evaluate patient satisfaction and the efficacy of home whitening with 10% carbamide peroxide in masking white spot lesions, as well as the presence of sensitivity and gingival irritation.

DETAILED DESCRIPTION:
The clinical trial aims to evaluate patient satisfaction and the efficacy of home whitening with 10% carbamide peroxide in masking white spot lesions, as well as the presence of sensitivity and gingival irritation. Patients with at least one white spot due to enamel development defects in any of the anterior teeth will be selected, up to a minimum of 67 lesions. An initial characterisation of the white spot lesions will be performed using different standardised photographs with cross-polarisation filters, fluorescence and transillumination. In addition, mapping will be performed using a spectrophotometer to record the L*a*b* parameters in the lesions and surrounding tissue, and patients will initially respond to a survey on their satisfaction with the lesions (VAS scale) and their impact on psychosocial well-being and oral health-related quality of life (PIDAQ and OHIP-14, respectively). Patients classified for the study will be whitened with 10% carbamide peroxide for 3 hours a day for 4 weeks, or until the desaturation obtained is to their liking, or until the CIELAB L* parameter measurements indicate stabilisation of brightness using the spectrophotometer. During treatment, the presence of sensitivity and irritation will be recorded using a VAS scale. Patients will be reviewed 4 weeks after the end of treatment and will respond again to the questionnaire on satisfaction, psychosocial impact of dental aesthetics and oral quality of life (PIDAQ and OHIP-14), and the lesions will be characterised again. The data obtained on satisfaction, PIDAQ and OHIP-14 surveys will be statistically analysed, as will the colour difference between the lesions and the surrounding tissue enamel at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age.
* Have white spots on teeth between 1.3 and 2.3 or between 3.3 and 4.3.
* No previous dental treatment on teeth affected by hypomineralisation lesions.
* No active caries lesions at any ICDAS II stage on the anterior teeth.
* Patients with satisfactory oral hygiene and periodontal health, who are not undergoing periodontal maintenance and who do not use chlorhexidine mouthwashes. Patients with recessions without sensitivity are included.

Exclusion Criteria:

* Patients who have previously undergone whitening treatment (less than 5 years ago).
* Patients undergoing orthodontic treatment.
* Patients with a history of trauma to the front teeth.
* Patients with endodontically treated anterior teeth.
* Pregnant or breastfeeding patients.
* Patients who smoke.
* Patients with periodontal disease.
* Patients with poor oral hygiene.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Degree of satisfaction with whitening on white spot lesions | 2 weeks
  The patient will answer questions using the PIDAQ questionnaire to assess whether they consider their white spot lesions to be masked after the whitening treatment.

SECONDARY OUTCOMES:
Effectiveness of masking white spot lesions | 2 weeks
  The lesions will be characterised as described above at 4 weeks and one month after the end of the whitening treatment. If the whitening treatment is prolonged, this will also be done at the end of the treatment. The effectiveness of masking will be determined by the colour difference between the lesions and the surrounding tissue using the CIELAB formula (De L'Eclairage, 1978):
  ∆Eab = [(∆L*)2 + (∆a*)2 + (∆b*)2]1/2. By definition, a tooth is considered masked when the colour difference (ΔEab) between the lesions and the surrounding healthy enamel is ΔEab ≤3.7, and unmasked if ΔEab > 3.7. A colour difference below the acceptability threshold of 3.7 was chosen as an indicator of masking.
  In addition, the colour change will also be calculated using the CIEDE 2000 formula:
  Additionally, the CIEDE2000 formula will be applied;
  ∆E00 = [(ΔL/kLSL)2 + (ΔC/kCSC)2 + (ΔH/kHSH)2 + RT(ΔC*ΔH/SC*SH)]1/2
  and the whiteness index (WI)
EVALUATION OF DENTAL SENSITIVITY | 2 weeks
  We will assess sensitivity and intensity using a visual analogue scale (VAS) from 0 to 10. Each patient will be given a diary covering the two weeks between appointments, which they will have to fill in daily. Zero will represent 'no pain' on the visual analogue scale and ten will represent 'severe pain'. Patients will be asked to record the worst result once a day, even if there has been no pain, marking with a vertical line the value corresponding to the intensity of their tooth sensitivity, which will then be measured in centimetres. If the patient marks any value above zero, it will be interpreted as tooth sensitivity. In cases of severe sensitivity, desensitising agents or analgesics/anti-inflammatories will be dispensed.
EVALUATION OF GINGIVAL IRRITATION | 2 weeks
  We will assess gingival irritation and the intensity of said irritation using a visual analogue scale (VAS) from 0 to 10 by means of a diary that will be provided together with the dental sensitivity diary, which the patient will fill in the same way, with zero being 'no gingival irritation' and ten being 'severe irritation'. Patients will be asked to record the worst result once a day, even if there has been no irritation, marking with a vertical line the value corresponding to the intensity of gingival irritation, which will then be measured in cm.
EVALUATION OF THE APPEARANCE OF NEW SPOTS | 2 weeks
  We will assess the appearance of new lesions during treatment using a visual analogue scale (VAS) from 0 to 10 in a diary that will be provided along with the tooth sensitivity diary, which the patient will fill out in the same way, with zero being 'very dissatisfied' and ten being 'very satisfied'. Patients will be asked to record the worst result once a day by marking with a vertical line the value corresponding to the intensity of gingival irritation, which will then be measured in centimetres.

CONTACTS AND LOCATIONS:
Overall Officials: Mª VICTORIA FUENTES, PhD Proffesor, Study Director — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided